CLINICAL TRIAL: NCT02202421
Title: Targeted Applied Behavior Analysis (T-ABA) Group Based Early Intervention for Parents of Children With Autism Spectrum Disorder (ASD)
Brief Title: T-ABA Group Based Early Intervention For Parents of Children With ASD
Acronym: T-ABA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI and study coordinator both left the institution.
Sponsor: The Cleveland Clinic (Other)
Collaborators: O'Neill Foundation (Unknown); CVS Caremark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCF IRB 14-429
Record Dates: First submitted 2014-07-22; First posted 2014-07-29 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Autism
Keywords: Autism; Applied Behavior Analysis
MeSH Terms: conditions — Autistic Disorder | interventions — tyrosine-4-azobenzenearsonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-ABA Parent Training Only (Active Comparator): Participants in the T-ABA Parent Training Only group will be given Targeted Applied Behavior Analysis (T-ABA) Intervention with five weeks of parent group training and five weeks of parent-therapists one-on-one sessions. They will also be offered eight one hour individual therapist-child applied behavior analysis sessions at the conclusion of the study if desired.
  Interventions: Behavioral: Targeted Applied Behavior Analysis (T-ABA)
- T-ABA Parent Group + Individual Therapy (Experimental): Participants in the T-ABA Parent Group plus Individual Therapy group will be given Targeted Applied Behavior Analysis (T-ABA) Intervention with five weeks of parent group training and five weeks of parent-therapists one-on-one sessions. They will also be offered eight one-hour individual therapist-child applied behavior analysis therapy sessions concurrent with the parent group and parent-therapist sessions.
  Interventions: Behavioral: Targeted Applied Behavior Analysis (T-ABA)

INTERVENTIONS:
Behavioral: Targeted Applied Behavior Analysis (T-ABA) — Participants will be enrolled in a five week Targeted Applied Behavior Analysis (T-ABA) parent therapy group. T-ABA parent groups will be 1.5 hours in length. Following the five weeks of parent group sessions, parents will participate in five weekly one-hour parent-therapist sessions in which a therapist will work one-on-one with the parent and their child. One treatment group (T-ABA Parent Group plus Individual Therapy) will also receive eight one-hour individual therapist-child applied behavior analysis therapy sessions concurrent with the parent group and parent-therapist sessions. The second treatment group (T-ABA Parent Training Only) will be offered eight one hour individual therapist-child applied behavior analysis sessions at the conclusion of the study if desired.

SUMMARY:
This study is a 10-week, randomized, parallel groups design which will evaluate the efficacy of T-ABA with combined parent training and individual child sessions versus T-ABA with individual sessions alone. T-ABA refers to Targeted Applied Behavior Analysis treatment, a form of behavior therapy used to promote skill development and reduce disruptive behavior in individuals with autism. Four key outcome assessment points will be used: baseline (week 0), midpoint (week 5), end-of-study (week 10), and follow-up (week 20). Participants receiving T-ABA parent training only will be offered eight individual therapy sessions at the end of the study. Total study participation is estimated to be ~ 10 weeks with a single follow-up assessment.

DETAILED DESCRIPTION:
This is a ten week study. The child will be randomized to one of two treatment groups. Assignment is chosen by chance (like flipping a coin). The two treatment groups are T-ABA (Targeted Applied Behavior Analysis) with parent training and T-ABA with parent training and individual child sessions. For both groups, study procedures will be the same except the T-ABA with parent training and individual child sessions group will receive eight one-to-one Applied Behavior Analysis (ABA) individual therapy sessions during the course of the study. Participants in the T-ABA with parent training group will be offered eight one-to-one ABA individual therapy sessions at the conclusion of the study.

During the child's participation in this study families are asked to not make any changes to his or her current neuropsychiatric medications or therapy for two weeks before the study begins and during his or her ten week participation. Medication changes may include increasing or decreasing the dose you receive, changing the time of day the child takes medication, starting a new medication, or discontinuing a current medication. Therapy the child receives may include speech, OT, PT, counseling, play therapy, music therapy, social skills training, special education services, socialization, recreational sports, or nutritional interventions. Therapy changes may include increasing or decreasing how often the child receives therapy, changing who the child receives therapy from, beginning a new therapy or discontinuing a current therapy.

The child will be asked to complete assessments before the start of the study. The child will complete a language assessment and an eye tracking task that will measure his or her attention to different pictures and videos. Families will complete questionnaires that examine the child's medical and family history as well as his or her current symptoms, functioning, and quality of life and families will be given a language collection device. This is like a recorder that will record every time the family or the child talks. Families will place the language collection device in the pocket of the child's clothing and it will record the language environment for two days. Families will return the language collection device to us. To help us better understand your child's medical condition, we will access the child's medical records to collect any previous evaluations and diagnoses.

During weeks 1 through 4, families will attend a parent training group. Each group will be 1.5 hours long and will focus on topics such as discrete trial teaching (breaking skills into small components in order to teach new information to the child), natural environment teaching (using the environment to increase the child's motivation to communicate), assessing and treating challenging behavior, using visual supports and teaching everyday living activities such as drinking from a cup or washing hands. During these groups families will have the opportunity to view examples and practice using the skills discussed.

During week 5, families will attend a parent training group. Families and their children will also be observed and videotaped by study staff for 10 minutes during which they will be asked to use the techniques you learned during the parent group. The video tape will be kept in the child's study file and will only be viewed by study staff as part of the research study. Families will also complete questionnaires that examine the child's medical and family history as well as his or her current symptoms, functioning, and quality of life and will be given a language collection device (like a tape recorder). They will place the language collection device in the pocket of the child's clothing and it will record his or her language and language environment for 2 days. They will return the language collection device to us.

During weeks 6 through 9 families and their children will attend a one-hour weekly parent-therapist session with a study staff member. They will practice using the techniques from the parent group with their child and the study staff member will provide them with coaching and feedback. Families can also bring along specific questions they have.

During week 10, families will attend a parent-therapist session. Families and their children will also be observed and videotaped by study staff for 10 minutes during which they will practice using the techniques from the parent group with their child. They will also complete questionnaires that examine the child's current symptoms, functioning, and quality of life and they will be given a language collection device. They will place the language collection device in the pocket of the child's clothing and it will record his or her language and language environment for 2 days. Families will return the language collection device to us. The child will also complete testing with a study staff. Testing will measure the child's language and attention to pictures and videos during an eye tracking task.

Ten weeks after the study is complete, families and their children will complete the same assessment procedures that were completed during week 10 in order to measure any changes that occurred after the end of the study.

If a family is in the T-ABA with parent training and individual child sessions group, the child will also receive one-to-one ABA therapy sessions during weeks 1 through 4 and 6 through 9. During the one-to-one ABA therapy sessions the child may work with the therapist on skills such as making eye contact when his or her name is called, playing with toys, asking for favorite foods or activities using words or gestures, making choices, taking turns or responding to one-step commands. Study staff will work with families to select programming to be completed with their child during these sessions.

If a family is in the T-ABA with parent training group, they will be asked if they'd like to schedule eight one-to-one ABA therapy sessions at the conclusion of the study (after follow-up assessments have been collected).

Families will receive assessment results in a brief report provided after testing is completed at visits 1, 5, 10 and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical DSM-5 diagnosis of Autism Spectrum Disorder (299.00).
* Age 2.0 (24 months) to 5.99 (71 months) at time of consent.
* If participant is using neuropsychiatric medication and/or receiving therapy (PT, OT, speech, ABA, etc.), these must be stable two weeks prior to their study participation and throughout the 10 week study period.

Exclusion Criteria:

* Age less than 2.0 (24 months) or greater than 5.99 (71 months) at time of consent.
* Individuals for whom neuropsychiatric medication (dose, dosing schedule, introduction of new medication, discontinuing current medication) or therapy (frequency of intervention, provider, introduction of new therapy, discontinuing current therapy) changes may occur two weeks prior to study or during the 10 week study period.
* Any participant who has previously received Applied Behavior Analysis (ABA) therapy (any form).
* Parent and/or guardian unable to speak, read and/or understand English.

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Increase in child utterances | 10 weeks
  The primary objective of this study is to determine whether T-ABA with parent training and individual child sessions is superior to T-ABA with parent training alone in improving child utterances as calculated by the LENA digital language processor.

SECONDARY OUTCOMES:
Child communication | 10 weeks
  To evaluate if T-ABA with combined child sessions and parent training is superior to T-ABA with parent training alone in increasing the number of child utterances as measured using the LENA Pro language collection device.
Autism and other behavioral symptoms | 10 weeks
  To evaluate if T-ABA with combined child sessions and parent training is superior to T-ABA with parent training alone in improving autism and other behavioral symptoms.
Language Scores | 10 weeks
  To evaluate if T-ABA with combined child sessions and parent training is superior to T-ABA with parent training alone in improving language scores on cognitive testing.
Adaptive Behavior | 10 weeks
  To evaluate if T-ABA with combined child sessions and parent training is superior to T-ABA with parent training alone in improving adaptive behavior.
Eye Tracking | 10 weeks
  To evaluate if T-ABA with combined child sessions and parent training is superior to T-ABA with parent training alone in improving eye tracking of social targets.
Global Functioning | 10 weeks
  To evaluate if T-ABA with combined child sessions and parent training is superior to T-ABA with parent training alone in improving global functioning via VB-MAPP.
Quality of Life | 10 weeks
  To evaluate if T-ABA with combined child sessions and parent training is superior to T-ABA with parent training alone in improving quality of life.

OTHER OUTCOMES:
Demographics and Clinical Variables | 10 weeks
  To evaluate whether baseline demographic and clinical variables (age, sex, IQ, parent education, parent occupation level, presence of a genetic syndrome) significantly predict patient outcomes.
Parent Fidelity | 10 weeks
  To assess if parent fidelity of T-ABA treatment predicts greater improvement in outcomes.
Parent Education | 10 weeks
  To evaluate parents' increased understanding of autism and strategies to manage their child's behavior, evaluated by a pre-/post-test regarding autism and therapeutic options.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Frazier, PhD, Principal Investigator — Cleveland Clinic Center for Autism
Locations (1):
- Cleveland Clinic Center for Autism, Cleveland, Ohio, United States

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders. Fifth ed. Arlington, VA: American Psychiatric Association; 2013.
- [Background] Kohler, F.W. Examining the services received by young children with autism and their families: A survey of parent responses. Focus on Autism and Other Developmental Disabilities. 1999;14:150-158.
- [Background] Stoner JB, Bock SJ, Thompson JR, Angell ME, Heyl BS, Crowley EP. Welcome to our world: Parent perceptions of interactions between parents of young children with ASD and educational professionals. Focus on Autism and Other Developmental Disabilities. 2005;20:39-51.
- [Background] Kogan MD, Strickland BB, Blumberg SJ, Singh GK, Perrin JM, van Dyck PC. A national profile of the health care experiences and family impact of autism spectrum disorder among children in the United States, 2005-2006. Pediatrics. 2008 Dec;122(6):e1149-58. doi: 10.1542/peds.2008-1057. PMID 19047216
- [Background] Minjarez MB, Williams SE, Mercier EM, Hardan AY. Pivotal response group treatment program for parents of children with autism. J Autism Dev Disord. 2011 Jan;41(1):92-101. doi: 10.1007/s10803-010-1027-6. PMID 20440638
- [Background] Coolican J, Smith IM, Bryson SE. Brief parent training in pivotal response treatment for preschoolers with autism. J Child Psychol Psychiatry. 2010 Dec;51(12):1321-30. doi: 10.1111/j.1469-7610.2010.02326.x. PMID 21073457